CLINICAL TRIAL: NCT05885126
Title: The Effect of Mandala Technique on Acute Nausea-vomiting and Comfort Level in Cancer Patients Receiving Outpatient Chemotherapy
Brief Title: The Effect of Mandala Technique on Acute Nausea-vomiting and Comfort Level in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Özlem KARDAŞ KİN, Nurse, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 123456123456
Record Dates: First submitted 2023-04-26; First posted 2023-06-01 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Chemotherapy-induced Nausea and Vomiting; Nursing Caries
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Intervention Model Description: The sample recruited for the research consisted of 38 individuals (19 individuals in the control group, 19 in intervention group) who were 18 years and older, were receiving a high emetogenic chemotherapy regimen for the first time, had sufficient fine motor skills to paint and were volunteering to participate in research. Exclusion criteria were any physical or mental disability that limited communication or coloring the mandala template. Homogeneity was ensured by including patients who received chemotherapy regimen with high emetogenicity. Patient lists numbered according to even and odd numbers were given in a sealed envelope to a practitioner independent from the researchers.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients in the intervention group were allowed to paint mandala templates for 30 minutes during chemotherapy treatment after premedication. Before the application, the patients were informed by the practitioner and given a laptop table, mandala coloring books and crayons, they were asked to paint a mandala template of their choice. The ambient light and the position of the laptop table were adjusted appropriately during the intervention to help the participants move freely and eliminate the environmental stimulus. In addition, there was no communication between the patient and the practitioner during the application. The patients in the intervention group were given the materials necessary for painting medallions after the treatment, and they were asked to apply at home for at least 30 minutes the day after the treatment. The patients were supported by telephone to paint while they were at home.
  Interventions: Other: MANDALA TECHNIQUE
- Control Group (No Intervention): Participants in the control group did not receive any intervention during or after treatment.

INTERVENTIONS:
Other: MANDALA TECHNIQUE — The ambient light and the position of the laptop table were adjusted appropriately during the intervention to help the participants move freely and eliminate the environmental stimulus. In addition, there was no communication between the patient and the practitioner during the application.
  Arms: Intervention Group

SUMMARY:
Cancer is an important health problem in the world and in our country, and it ranks second among the causes of death in our country (20.7%). Chemotherapy, one of the most commonly used methods in cancer treatment, causes many physical and emotional symptoms while treating the disease. Nausea-vomiting is a common problem in cancer care, especially in patients receiving chemotherapy.

In the literature, there are studies examining non-pharmacological interventions for the prevention and management of nausea and vomiting in patients receiving chemotherapy, and it is seen that the interventions are mostly within the scope of complementary and alternative approaches. Patients receiving ambulatory chemotherapy may experience anticipatory nausea in particular, and this is likely to affect the individual's comfort level. In studies conducted in the field, the comfort level of cancer patients receiving chemotherapy was determined as moderate.

Today, mandalas are used effectively in the field of art therapy. The possibility of using mandala in all age groups has contributed to the treatment process of different diseases and disorders, and its effectiveness has been presented to the scientific world with many researches around the world. In adults, the mandala has been used both in the treatment of psychiatric disorders and as a tool to observe the effects of treatments. Art therapy including mandala drawing has significantly reduced the severity of trauma symptoms in individuals with anxiety disorders and post-traumatic stress disorder. In the study of Zhao & Tang (2017) it was determined that mandala drawing therapy reduced the anxiety of cancer patients.

If the reduction of nausea-vomiting affects the comfort level and the person is relieved, a more effective treatment environment is created and the quality of life of the person is increased. In the literature, very limited studies have been reached on the use of the mandala drawing technique in cancer patients. National and international research examining the mandala drawing technique, especially in patients receiving ambulatory chemotherapy, could not be reached. The aim of this study is to determine the effect of mandala drawing technique on nausea-vomiting and comfort level in patients receiving ambulatory chemotherapy. It is anticipated that the study to be conducted will contribute to nursing interventions in the cancer care process and lead to the planning of new research on the subject.

DETAILED DESCRIPTION:
This research was planned in a quasi-experimental design with pretest-posttest control group. It is aimed to determine the effect of mandala technique on nausea-vomiting and comfort level in patients receiving ambulatory chemotherapy.

For this purpose, the research will be carried out with cancer patients receiving chemotherapy treatment on an outpatient basis at Gaziantep University Medical Faculty Training and Research Hospital and Gaziantep University Oncology Hospital between December 2022 and April 2023. The population of my research will consist of patients who receive outpatient chemotherapy treatment at Gaziantep University Faculty of Medicine Oncology Hospital. Individuals who meet the sampling selection criteria from the specified universe will constitute the sample of the research. Experimental research requires at least 20 samples. In order for a test to meet the parametric test conditions, references were made to the sources stating that the groups must have at least 30 individuals. In the research group of our study, it was planned to include 30 application and 30 control group patients. When these numbers are reached, it is planned to determine the sample impact power by performing power analysis, and to terminate the research when at least 80% preferably 100% positive impact power is reached. Randomization of the sample will be achieved by accepting the first patient who applied to the outpatient chemotherapy unit randomly and with an appointment at the beginning of the study to the control group, and the next patient to the experimental group. The patients will be included in the experimental and control groups in this order until the sample size is reached.

The implementation of the study will start after the necessary permissions are obtained, and the application group will be asked to paint the mandalas provided by the researcher for at least 30 minutes while they are in the chemotherapy unit. The patients will be given the necessary materials during their stay at home, they will be asked to paint mandalas at home for 4 days, and the patient will be supported by phone. No treatment other than standard care will be performed for the control group.

ELIGIBILITY:
Inclusion criteria for the research:

* 18 years of age or older, conscious, literate, not having vision and hearing problems, being able to communicate verbally,
* Receiving outpatient chemotherapy treatment at Gaziantep University Faculty of Medicine Training and Research Hospital and Gaziantep University Oncology Hospital,
* Receiving a medium and high emetogenic effective chemotherapy regimen
* Having sufficient fine motor skills to paint,
* Not having any diagnosed psychiatric disorder,
* Agreeing to participate in the research

Exclusion criteria from the study:

* Having any communication problems,
* Having sufficient fine motor skills to paint,
* Refusal to participate in the research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Acute Nausea-Vomiting | 5 months
  The change in the patient's nausea and vomiting will be observed using The MASCC Antiemesis Tool (MAT)
Genel Comfort Level | 5 months
  The change in the patient's comfort level will be observed by using the General Comfort Scale Short Form.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem KARDAŞ KİN, Principal Investigator — Gaziantep Islamic and Technology University
Locations (2):
- Turkey (Türkiye) (2):
  - Gaziantep Islamic and Technology University, Pazarcık, Kahramanmaraş
  - Gaziantep İslamic and Technology University, Gaziantep

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Celik A, Kin OK. Clinical Trial of Mandala Coloring for Management of Chemotherapy-Induced Nausea and Vomiting. Altern Ther Health Med. 2024 Dec;30(12):13-17. PMID 39565703